CLINICAL TRIAL: NCT06020326
Title: A Retrospective Cohort Study of Hemorrhagic Fever With Renal Syndrome
Brief Title: A Retrospective Cohort Study of HFRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qin Ning, Director, Department of Infection, Tongji Hospital
Other Study IDs: REHEAL
Record Dates: First submitted 2023-08-17; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-07

CONDITIONS: HFRS
MeSH Terms: conditions — Hemorrhagic Fever with Renal Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this retrospective cohort study is to learn about the clinial characteristics of HFRS patients, explore the risk factors of the occurrence and death of HFRS, and build a risk prediction model for HFRS.

DETAILED DESCRIPTION:
HFRS remains an important public health issue in China, which not only poses a threat to people's physical health and safety, but also has a serious impact on social and economic development. At present, there is no unified standard for clinical prediction of the occurrence and death of HFRS. In order to better prevent and treat HFRS, this multicenter retrospective clinical study is designed to include HFRS inpatients, and collect their demographics, epidemiological history, hospitalization information, clinical manifestation, laboratory results, imaging results, treatment plan and outcome.

ELIGIBILITY:
Inclusion Criteria:

The patients must meet all of the following criteria:

* Inpatient with clinical diagnosis of Haemorrhagic Fever with Renal Syndrome

Exclusion Criteria:

Exclude patients who meet any of the following criteria:

* Patients with previous chronic kidney disease
* Pregnant or perinatal patients
* Patients unsuitable for inclusion by investigators' evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with HFRS diagnosed
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
short-term mortality | 90 days post diagnosed HFRS
  28-day and 90-day mortality after diagnosed as HFRS

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Professor, Principal Investigator — Tongji Hospital
Locations (8):
- China (8):
  - No.1 Peoples Hospital of Guangshui, Guangshui, Hubei
  - Huanggang Central Hospital, Huanggang, Hubei
  - People's Hospital of Luotian County, Huanggang, Hubei
  - People's Hospital of Macheng City, Affiliated Hospital of Hubei University of Science and Technology, Macheng, Hubei
  - Qianjiang Central Hospital, Qianjiang, Hubei
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science & Technology, Wuhan, Hubei
  - Xianning Central Hospital, Xianning, Hubei
  - The Third Peoples Hospital of Yichang, Yichang, Hubei